CLINICAL TRIAL: NCT05321095
Title: Screening for Albuminuria at the First Line for Early Identification of Chronic Kidney Disease: a Pilot Study
Brief Title: Screening for Albuminuria at the First Line for Early Identification of CKD
Acronym: SALINE
Status: Completed | Type: Observational
Sponsor: General Practitioners Research Institute (Network)
Collaborators: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: GPRI-21004-CKD
Record Dates: First submitted 2022-02-07; First posted 2022-04-11 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-02

CONDITIONS: Chronic Kidney Diseases; Albuminuria
MeSH Terms: conditions — Renal Insufficiency, Chronic; Albuminuria

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Screening: Only one group will be evaluated during the SALINE study. Everyone that meets the inclusion criteria of having a high risk for albuminuria is invited to participate. During participation, subjects are asked to collect one or more urine samples for albuminuria determination. If albuminuria is high (>= 3,0 mg/mmol) subjects are invited for a visit. During the visit non-invasive measurements (BMI, PoC HbA1c, eGFR, blood pressure and heart rate) are taken to determine the cardiovascular risk. Furthermore, medication use is reviewed.
  Interventions: Diagnostic Test: Albuminuria test; Diagnostic Test: HbA1c test; Diagnostic Test: Creatinine test

INTERVENTIONS:
Diagnostic Test: Albuminuria test — During participation, subjects are asked to collect one or more urine samples for albuminuria determination.
  Other Names: PeeSpot
Diagnostic Test: HbA1c test — During the screening visit, HbA1c will be measured with a point-of-care test (Affinion HbA1c, Abbott).
  Other Names: Affinion HbA1c
Diagnostic Test: Creatinine test — During the screening visit, creatinine will be measured with a point-of-care test (i-STAT Alinity handheld analyser, Abbott).
  Other Names: i-STAT Alinity

SUMMARY:
Early detection of kidney disease

DETAILED DESCRIPTION:
Early detection and appropriate treatment of kidney disease is important as this may prevent future cardiovascular complications and end-organ damage more effectively than intervention in more advanced stages of disease. There is a well-established relationship between albuminuria and renal- and cardiovascular disease. Elevated albuminuria has a relatively high prevalence in the general population (5-9%). The prevalence of albuminuria is even higher in high-risk patients with diabetes Mellitus, hypertension, obesity, cardiovascular disease and lipid disorders. Adequate treatment of albuminuria, preferable at early stages can prevent both cardiovascular and renal disease progression. However, scarce epidemiological data show that albuminuria measurements are only conducted in a minority of individuals and disease recognition is suboptimal, even in high-risk groups. The current study aims to evaluate if and how early identification of chronic kidney disease by targeted screening of albuminuria levels is feasible in primary care (pharmacies and general practitioners) to optimally discover and treat patients with elevated albuminuria.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Mellitus (diagnosis or prescription for the disease based on the NHG guidelines)
* Adipositas (diagnosis)
* Hypertension (diagnosis or prescription for the disease based on the NHG guidelines)
* Cardiovascular disease (diagnosis, specified in protocol section 5.2.2)
* Lipid disorder (diagnosis or prescription for the disease based on the NHG guidelines)

Exclusion Criteria:

* Inability to understand and sign the informed consent form
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a high risk of (developing) chronic kidney disease will be recruited in primary care practices and pharmacies from the General Practitioners Research Institute (GPRI) network. The organizational model of GPRI is based on the participation of independent practices and pharmacies in the Netherlands, well-trained GPs, pharmacists and their staff. Male and female subjects aged above 18 years that meet the inclusion criteria will be eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
The prevalence of elevated albuminuria | 1-2 weeks after invitation
  defined as a confirmed urinary albumin creatinine ratio (UACR) ≥ 3.0 mg/mmol.

SECONDARY OUTCOMES:
The prevalence of unknown elevated albuminuria | through study completion, an average of 5 weeks
  defined as elevated albuminuria not reported by the subject or previously recorded in electronic medical records of the subjects' general practice or pharmacy.
Average costs per subject | through study completion, an average of 5 weeks
  by screening for albuminuria via pharmacies versus general practitioners.
the proportion of invited subjects that was identified as having hidden kidney disease | through study completion, an average of 5 weeks
  by screening for albuminuria via pharmacies versus general practitioners.

CONTACTS AND LOCATIONS:
Overall Officials: H.J. Lambers Heerpink, Prof. dr., Principal Investigator — University Medical Center Groningen
Locations (1):
- General Practitioners Research Institute, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van Mil D, Kieneker LM, Harms E, Prins GH, van Geer-Postmus I, Mepschen M, Leving MT, Stoker N, Herman Kocks JW, Gansevoort RT, Lambers Heerspink HJ. Effectiveness of a systematic home-based albuminuria screening programme to detect chronic kidney disease in high-risk individuals in primary care (SALINE): a cross-sectional screening study. EClinicalMedicine. 2025 Apr 8;82:103185. doi: 10.1016/j.eclinm.2025.103185. eCollection 2025 Apr. PMID 40247889